CLINICAL TRIAL: NCT03972852
Title: Establishment of an Anaesthetic Protocol for Examinations Under Anaesthesia for Children With Glaucoma or Suspected Glaucoma - Correlation of Bispectral Index (BIS) and Intraocular Pressure (IOP)
Brief Title: Establishment of an Anaesthetic Protocol for Examinations for Children With Glaucoma or Suspected Glaucoma
Acronym: eyeBIS
Status: Completed | Type: Observational
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Nina Pirlich, Dr. med., Principle Investigator, Johannes Gutenberg University Mainz
Other Study IDs: eyeBIS 1.0
Record Dates: First submitted 2019-05-31; First posted 2019-06-04 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Anesthesia; Intraocular Pressure; Glaucoma, Suspect; Pediatric Glaucoma
MeSH Terms: conditions — Ocular Hypertension; Hydrophthalmos

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Correct measurement of the intraocular pressure of children with glaucoma or suspected glaucoma is essential for diagnosis and therapy.

Despite new non-invasive measurement methods most of the children are uncooperative during the ophthalmological examination. Therefore examination under anaesthesia is needed.

A lot of perioperative factors influence the measurement of intraocular pressure.

Established and safe anaesthetic regimes have been modified regarding these factors. Aim of the study is to evaluate, if a standardized anaesthetic protocol generates reliable and reproducible measured values.

ELIGIBILITY:
Inclusion Criteria:

* Indication for a general anesthesia (laryngeal mask) and ophthalmological examination and probably surgery
* Children with glaucoma or suspected glaucoma
* ASA classification I-III
* written informed consent of the legal representatives

Exclusion Criteria:

* Contraindication for a laryngeal mask airway
* Known allergy to propofol or remifentanil

Ages: 5 Months to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with glaucoma or suspected glaucoma for ophthalmological examination or surgery
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2025-12-28 (Actual)

PRIMARY OUTCOMES:
Correlation of depth of anesthesia an intraocular pressure | 1 day
  The primary outcome measure is the association between intraocular pressure and bispectral index.

SECONDARY OUTCOMES:
Bland Altmann Correlation of Applanation tonometry and rebound tonometry | 1 day
  Comparison of two different examination tools
Normal range of pediatric intraocular pressure | 1 day
  Defining the normal range of pediatric intraocular pressure
Correlation of the corneal thickness and the intraocular pressure | 1 day
  Regression

CONTACTS AND LOCATIONS:
Locations (1):
- Johannes Gutenberg - Universität, Mainz, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pirlich N, Grehn F, Mohnke K, Maucher K, Schuster A, Wittenmeier E, Schmidtmann I, Hoffmann EM. Anaesthetic protocol for paediatric glaucoma examinations: the prospective EyeBIS Study protocol. BMJ Open. 2021 Oct 5;11(10):e045906. doi: 10.1136/bmjopen-2020-045906. PMID 34610927